CLINICAL TRIAL: NCT02270099
Title: Clinical Evaluation of the Aptima® Herpes Simplex Viruses 1 & 2 Assay on the Panther® System in Swab Specimens From Symptomatic Subjects Presenting With a Suspected Herpes Lesion(s)
Brief Title: Evaluation of the HSV 1 & 2 Assay in Specimens From Symptomatic Subjects
Status: Completed | Type: Observational
Sponsor: Hologic, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: A10921-HSVPS-CSP-01
Record Dates: First submitted 2014-10-16; First posted 2014-10-21 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Herpes Simplex Infections
MeSH Terms: conditions — Herpes Simplex

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — lesion swab
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects with suspected HSV Lesions

SUMMARY:
This clinical performance study is being conducted to evaluate the performance of the Aptima Herpes Simplex Viruses 1 & 2 assay for detection of herpes simplex virus (HSV) type 1 (HSV-1) and HSV type 2 (HSV-2) in swab samples prospectively collected from suspected HSV lesions. Specimens collected using swabs from viral transport medium (VTM)collection kits and Aptima swab collection kits will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* The subject has at least 1 active lesion (lesion with exudates and cellular material; eg, vesicle, ulcer) that is suspected to be caused by HSV (as determined by the clinician)
* The subject and/or legally authorized representative is willing and able to provide consent prior to study participation (a minor will need the documented consent of his/her parent or legal guardian, unless the site has an institutional review board-approved waiver for parental consent for minors)

Exclusion Criteria:

* The subject has only HSV lesions without exudates and cellular material
* The subject used a topical or oral antiviral medication used to treat HSV within 21 days of enrollment
* Subject already participated in this study
* Subject has a history of illness that the principal investigator (PI) or designee considers could interfere with or affect the conduct, results, and/or completion of the study
* Subject has a history of illness that the PI or designee considers could create an unacceptable risk to the subject if enrolled in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male and female subjects attending participating US collection sites and presenting with suspected HSV lesion(s) will be eligible for the study. Sites may include family planning, general practice, dermatology, research, sexually transmitted infection, adolescent, and public health clinics. There are no age restrictions for this study.
Sampling Method: Non-Probability Sample
Enrollment: 839 (Actual)
Dates: Start 2014-12; Primary Completion 2016-08 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of sensitivity and specificity of the Aptima HSV 1 & 2 Assay on Panther | 1 day
  Sensitivity and specificity of the Aptima HSV 1 & 2 assay will be determined by comparing assay results to results from a reference method representing the true infected status of the subjects. Sensitivity will be reported as the percentage of subjects with an HSV infection who test positive by the Aptima HSV 1 & 2 assay. Specificity will be reported as the percentage of subjects without an HSV infection who test negative by the Aptima HSV 1 & 2 assay.

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Ziermann, Study Director — Hologic, Inc.
Locations (22):
- United States (22):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Elite Clinical Studies, LLC, Phoenix, Arizona
  - Sherif Khamis MD, Inc, Canoga Park, California
  - Mills Clinical Research, Los Angeles, California
  - Planned Parenthood of the Rocky Mountains, Denver, Colorado
  - Yale School of Medicine, New Haven, Connecticut
  - Perimeter Institute for Clinical Research, Inc. (PICR Clinic), Atlanta, Georgia
  - Advanced Clinical Research, Boise, Idaho
  - Indiana University School of Medicine, Indianapolis, Indiana
  - LSU Health Science Center, New Orleans, Louisiana
  - LSU Health Science Center - Shreveport, Shreveport, Louisiana
  - IRC Clinics, Towson, Maryland
  - University of Mississippi Medical Center/Crossroads Clinic (MSDH), Jackson, Mississippi
  - Quality Clinical Research Inc., Omaha, Nebraska
  - Rochester Clinical Research, Inc., Rochester, New York
  - Laboratory Corporation of America, Burlington, North Carolina
  - Westover Heights Clinic, Portland, Oregon
  - Planned Parenthood of Southeastern Pennsylvania, Philadelphia, Pennsylvania
  - Geneuity Clinical Research Services, Maryville, Tennessee
  - Planned Parenthood Gulf Coast, Inc., Houston, Texas
  - Center for Clinical Studies, Webster, Texas
  - American Regional University Pathologists, Salt Lake City, Utah